CLINICAL TRIAL: NCT05161845
Title: A Phase IV Randomized, Blinded Clinical Trial to Assess Measles Mumps and Rubella Combined Vaccine, Live, (MMR) Lot-to-lot Consistency in Healthy Chinese Children at the Age of 8-12 Months
Brief Title: Clinical Trial of Measles, Mumps and Rubella Combined Vaccine, Live
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SIBP-MMR-01
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2021-12

CONDITIONS: Immunotoxicity; Vaccine
Keywords: MMR Combined Vaccines; safety; immunogenicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Participants randomized to receive one injections of 0.5 mL Measles, Mumps and Rubella Combined Vaccine, Live at Day 0.
  Interventions: Biological: Measles, Mumps and Rubella Combined Vaccine, Live

INTERVENTIONS:
Biological: Measles, Mumps and Rubella Combined Vaccine, Live — 0.5ml of reconstituted vaccine per container. 0.5 ml per single human dose containing not less than 3.0 lg CCID50 of both live measles virus and rubella virus and 4.3 lg CCID50 of live mumps virus.

SUMMARY:
To evaluate the immunogenicity, lot-to-lot consistency and safety of three consecutive batches of Measles, Mumps and Rubella Combined Vaccine, Live.

DETAILED DESCRIPTION:
To assess Measles Mumps and Rubella Combined Vaccine, Live, (MMR) lot-to-lot consistency in healthy Chinese Children at the age of 8-12 months, and the participants randomized to receive one injections of 0.5 mL Measles, Mumps and Rubella Combined Vaccine, Live at day 0.

ELIGIBILITY:
Inclusion Criteria:

Provide vaccination certificate and birth certificate for healthy children aged 8-12 months;

* Volunteers' legal guardian informed consent, volunteered to participate and signed an informed consent form；
* The volunteer's legal guardian has the ability to understand the research procedures, use the thermometer, scale and fill in the diary card as required, and can complete the clinical study in accordance with the requirements of the clinical trial protocol.

Exclusion Criteria:

* The axillary body temperature on the day of enrollment was more than 37.0 ℃;
* Have suffered from measles, mumps and rubella in the past or are suffering from measles, mumps and rubella;
* Any previous vaccination containing measles, mumps and rubella;
* Persons known to be allergic to any ingredient in the investigational vaccine;
* Any previous history of vaccine or drug allergy;
* Premature (delivered before the 37th week of pregnancy) and low weight (birth weight < 2500g);
* History of dystocia, asphyxia rescue and nervous system damage;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Acute disease, serious chronic disease or acute attack of chronic disease on the day of vaccination;
* Have a history of live attenuated vaccine within 28 days before vaccination and other vaccines within 7 days;
* Those who receive immune enhancement or inhibitor treatment within 3 months (continuous oral or drip for more than 14 days);
* Suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* History of asthma, unstable in the past two years, requiring emergency treatment, hospitalization, intubation, oral or intravenous corticosteroids;
* Have received blood or blood related products;
* Patients with progressive nervous system diseases have a history of convulsion, epilepsy, encephalopathy, GuillainBarre syndrome, mental history or family history;
* Have a history of abnormal coagulation function (such as coagulation factor deficiency and coagulation diseases);
* Plan to move out before the end of the study or leave for a long time during the scheduled study visit;
* Participating in or planning to participate in other clinical trials in the near future;
* The investigator judges any situation that is not suitable to participate in this clinical trial.

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1068 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The geometric mean concentrations (GMC) | 42 days
  GMC of measles, mumps and rubella antibodies should be compared 42 days after vaccination, and detected by enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
The positive conversion rate of antibodies | 42 days
  1. The positive conversion rate of antibodies to measles, mumps and rubella in each group 42 days after vaccination.The seroconversion rate refers to the proportion of subjects whose serum antibodies are negative before vaccination, which turn positive after vaccination, or serum antibodies are positive before vaccination, which increased by 4 times or more after vaccination.
The Seropositivity rate | 42 days
  The seroprevalence rate refers to the proportion of subjects whose serum antibodies are positive. The cut-off for seropositivity for the antibody titers is as follows:
  1. Anti-measles IgG antibody concentration by ELISA of >200 mIU/mL.
  2. Anti-mumps IgG antibody concentration by ELISA of >100 U/mL.
  3. Anti-rubella IgG antibody concentration by ELISA of >20 IU/mL
The incidence of adverse events within 14 days | 14 days
  The incidence of adverse events within 14 days after vaccination
All adverse events | 42 days
  All adverse events from day 0 to 42 after vaccination
Serious adverse events | 180 days
  Serious adverse events within 6 months after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No